CLINICAL TRIAL: NCT05036824
Title: Intensive Dose Tinzaparin in Hospitalized COVID19 Patients
Brief Title: Intensive Dose Tinzaparin in Hospitalized COVID-19 Patients
Acronym: INTERACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, K.Akinosoglou MD,PhD, Study Principal Investigator, University Hospital of Patras
Other Study IDs: 18634/23-7-2021 pend. aprooval
Record Dates: First submitted 2021-08-13; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Hospitalization
Keywords: SARS-CoV-2; Tinzaparin; LMWH; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tinzaparin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COVID-19 patients: Patients admitted to hospital with COVID-19, PCR+ SARS-CoV-2 infection administered thromboprophylaxis with tinzaparin.
  Dosage: intermediate or therapeutic dose Frequency of tinzaparin administration: once daily Duration: Unknown
  Interventions: Drug: tinzaparin

INTERVENTIONS:
Drug: tinzaparin — Daily tinzaparin administration: 8000 - 14000 Anti-Xa IU
  Other Names: Innohep

SUMMARY:
The primary objective of this study is to evaluate the current management approach with "intermediate" or "therapeutic" doses of tinzaparin for thromboprophylaxis in hospitalized patients, non on ICU organ support, with confirmed COVID-19.

DETAILED DESCRIPTION:
A prothrombotic state, attributable to a cytokine storm induced by severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2) and leading to activation of the coagulation cascade, is a recognized feature of Coronavirus disease 2019 (COVID-19) infection. This can manifest in venous thromboembolism (VTE), arterial thrombosis events (ATE), and disseminated intravenous coagulation (DIC) and coagulopathy are reflective of more severe disease and adverse prognosis. A significant number of patients with COVID-19 require single or multiple organ support on the Intensive Care Unit (ICU), estimated to be between 12 and 17% of patients. with the reported mortality in these cohorts between 25 and 40%.

International guidelines recommend that hospitalized patients with COVID-19 should receive pharmacological prophylaxis against VTE, in the absence of contraindications. With respect to how VTE prophylaxis is achieved, Low Molecular Weight Heparins (LMWH), in addition to their well-known anticoagulant properties, appear to have additional antiviral and anti-inflammatory effects that may be potentially beneficial in hospitalized COVID-19 patients.

Though international and national guidelines state that all hospitalized patients with COVID-19 should receive pharmacologic thromboprophylaxis, the rising incidence of thrombotic complications in COVID-19 patients has led a lot of hospitals to adopt the strategy of increasing the dose of anticoagulation for prophylaxis to 'intermediate' or "therapeutic" doses using a risk-adapted strategy with increased doses administration based on factors associated with increased risk; clinicians weigh the benefits and risks of therapeutic anticoagulation in terms of thrombosis and major bleeding risk for individual patients.

Additionally, LMWHs have different physicochemical characteristics as a result of the diverse methods of their manufacturing. The variations in molecular composition and pharmacological properties of LMWHs are reflected in differences in their clinical efficacy and safety. Each LMWH should, therefore, be considered as a unique substance. Tinzaparin is the only LMWH known that is prepared by enzymatic hydrolysis with heparinase. Due to its preparation method, tinzaparin has distinct properties than other LMWHs including and not limited to: higher Anti-IIa activity and Anti-Xa/Anti-IIa activity ratio, the higher release of Tissue Factor Pathway Inhibitor (TFPI), less dependence from renal function for its clearance, and more complete neutralization from its antidote, if needed. Due to the key role of increased Thrombin generation (IIa) and Tissue factor (TF) pathway activation in COVID-19-associated thrombosis , special properties of tinzaparin in Anti-IIa activity and TFPI production and release from endothelial cells, as well as significant effects of TFPI in various vascular, inflammatory, cardiovascular, hematological and oncological disorders, tinzaparin could have an expanded role beyond its well-known anticoagulant function.

The purpose of this study is to evaluate the overall clinical effectiveness and safety of 'intermediate' or "therapeutic" doses of anticoagulation with tinzaparin administered for thromboprophylaxis in COVID-19 patients with moderate disease severity during hospitalization in Greek hospitals.

ELIGIBILITY:
Inclusion Criteria

1. Patients admitted to hospital with COVID-19, PCR+ SARS-CoV-2 infection (from any specimen) administered thromboprophylaxis with tinzaparin in intermediate or therapeutic dose
2. Age ≥ 18 years
3. Signed informed consent

Exclusion Criteria

1. Patients admitted to ICU with COVID-19, PCR+ SARS-CoV-2 infection (from any specimen)
2. Age < 18 years
3. Pregnancy
4. Current diagnosis or suspicion of pulmonary thromboembolism or deep vein thrombosis
5. Progression to death was imminent and inevitable within 24 hours from the admission, irrespective of the provision of treatments
6. Not signed informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with COVID-19 infection administered thromboprophylaxis with tinzaparin
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of thrombotic events | through study completion, an average of 6 months
  Evaluate the incidence of thrombotic events: total & per type e.g. PE, DVT, symptomatic, incidental, proximal, distant etc. (Measured as percentage of events in relation to the study population)
Incidence of bleeding events | through study completion, an average of 6 months
  Evaluate τηε ιncidence of bleeding events (total & per type e.g. Major, CRNMB and minor) (Measured as percentage of events in relation to the study population)

SECONDARY OUTCOMES:
WHO progression scale | through study completion, an average of 6 months
  Evaluate the patients in relation to World Health Organization (WHO) progression scale (range from 0 (healthy) to 10 (death); values below or equal to 5 correspond to the absence of any oxygen supply beside nasal or facial mask).
Length of hospital stay | through study completion, an average of 6 months
  Evaluate the length of hospital stay (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Akinosoglou, MD,PhD, Principal Investigator — University Hospital of Patras
Locations (7):
- Greece (7):
  - University Hospital of Patras, Pátrai, Achaia
  - Evangelismos General Hospital, Athens, Attica
  - General Hopital Elpis, Athens, Attica
  - University General Hospital of Ioannina, Ioannina, Epirus
  - General Hospital of Kerkira "Ag. Irini", Corfu, Ionian Islands
  - General Hospital of Kozani "Mamatsio", Kozani, Macedonia
  - Genereal Hospital of Patras "Ag. Andreas", Patras, Peloponnese

IPD SHARING:
Plan to Share IPD: Undecided
Data can e available after publication of results to other researchers upon a reasonable request.

REFERENCES:
- [Background] Arachchillage DRJ, Laffan M. Abnormal coagulation parameters are associated with poor prognosis in patients with novel coronavirus pneumonia. J Thromb Haemost. 2020 May;18(5):1233-1234. doi: 10.1111/jth.14820. No abstract available. PMID 32291954
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Docherty AB, Harrison EM, Green CA, Hardwick HE, Pius R, Norman L, Holden KA, Read JM, Dondelinger F, Carson G, Merson L, Lee J, Plotkin D, Sigfrid L, Halpin S, Jackson C, Gamble C, Horby PW, Nguyen-Van-Tam JS, Ho A, Russell CD, Dunning J, Openshaw PJ, Baillie JK, Semple MG; ISARIC4C investigators. Features of 20 133 UK patients in hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: prospective observational cohort study. BMJ. 2020 May 22;369:m1985. doi: 10.1136/bmj.m1985. PMID 32444460
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Moores LK, Tritschler T, Brosnahan S, Carrier M, Collen JF, Doerschug K, Holley AB, Jimenez D, Le Gal G, Rali P, Wells P. Prevention, Diagnosis, and Treatment of VTE in Patients With Coronavirus Disease 2019: CHEST Guideline and Expert Panel Report. Chest. 2020 Sep;158(3):1143-1163. doi: 10.1016/j.chest.2020.05.559. Epub 2020 Jun 2. PMID 32502594
- [Background] Spyropoulos AC, Levy JH, Ageno W, Connors JM, Hunt BJ, Iba T, Levi M, Samama CM, Thachil J, Giannis D, Douketis JD; Subcommittee on Perioperative, Critical Care Thrombosis, Haemostasis of the Scientific, Standardization Committee of the International Society on Thrombosis and Haemostasis. Scientific and Standardization Committee communication: Clinical guidance on the diagnosis, prevention, and treatment of venous thromboembolism in hospitalized patients with COVID-19. J Thromb Haemost. 2020 Aug;18(8):1859-1865. doi: 10.1111/jth.14929. No abstract available. PMID 32459046
- [Background] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Background] Poterucha TJ, Libby P, Goldhaber SZ. More than an anticoagulant: Do heparins have direct anti-inflammatory effects? Thromb Haemost. 2017 Feb 28;117(3):437-444. doi: 10.1160/TH16-08-0620. Epub 2016 Dec 15. PMID 27975101
- [Background] Thachil J. The versatile heparin in COVID-19. J Thromb Haemost. 2020 May;18(5):1020-1022. doi: 10.1111/jth.14821. Epub 2020 Apr 27. No abstract available. PMID 32239799
- [Background] Fegan CD. Tinzaparin as an antithrombotic: an overview. Hosp Med. 1998 Feb;59(2):145-8. PMID 9797891
- [Background] Linhardt RJ, Gunay NS. Production and chemical processing of low molecular weight heparins. Semin Thromb Hemost. 1999;25 Suppl 3:5-16. PMID 10549711
- [Background] Matzsch T, Bergqvist D, Hedner U, Ostergaard P. Effects of an enzymatically depolymerized heparin as compared with conventional heparin in healthy volunteers. Thromb Haemost. 1987 Feb 3;57(1):97-101. PMID 3590085
- [Background] Padilla A, Gray E, Pepper DS, Barrowcliffe TW. Inhibition of thrombin generation by heparin and low molecular weight (LMW) heparins in the absence and presence of platelet factor 4 (PF4). Br J Haematol. 1992 Oct;82(2):406-13. doi: 10.1111/j.1365-2141.1992.tb06437.x. PMID 1329921
- [Background] McFadyen JD, Stevens H, Peter K. The Emerging Threat of (Micro)Thrombosis in COVID-19 and Its Therapeutic Implications. Circ Res. 2020 Jul 31;127(4):571-587. doi: 10.1161/CIRCRESAHA.120.317447. Epub 2020 Jun 26. PMID 32586214
- [Background] Bajaj MS, Bajaj SP. Tissue factor pathway inhibitor: potential therapeutic applications. Thromb Haemost. 1997 Jul;78(1):471-7. PMID 9198199
- [Background] Kaiser B, Hoppensteadt DA, Fareed J. Tissue factor pathway inhibitor: an update of potential implications in the treatment of cardiovascular disorders. Expert Opin Investig Drugs. 2001 Nov;10(11):1925-35. doi: 10.1517/13543784.10.11.1925. PMID 11772296
- [Background] Bochenek J, Puskulluoglu M, Krzemieniecki K. The antineoplastic effect of low-molecular-weight heparins - a literature review. Contemp Oncol (Pozn). 2013;17(1):6-13. doi: 10.5114/wo.2013.33766. Epub 2013 Mar 15. PMID 23788954

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT05036824/Prot_SAP_000.pdf